CLINICAL TRIAL: NCT00515307
Title: In-Vitro Transdifferentiation of Mesenchymal Stem Cells to Hepatocytes and Allogenic Transplantation of Hepatocytes to the Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Bone Marrow Stem Cells as a Source of Allogenic Hepatocyte Transplantation in Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Reza Malekzadeh, Digestive Disease Research Center, Medical Sciences/ University of Tehran
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDRC 85-15
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Hypercholesterolemia, Familial
Keywords: Hypercholesterolemia, Familial; Bone marrow; Mesenchymal stem cell; Hepatocyte
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Procedure: Cellular transplantation

INTERVENTIONS:
Procedure: Cellular transplantation — 600 million to 1 billion cells will be infused through the portal vein over 30 minutes. Infusion will be done one time.

SUMMARY:
Patients with homozygous familial hypercholesterolemia has very high serum cholesterol levels despite receiving lipid lowering drugs (e.g. statins, etc). Most of such patients die before the age of 20 due to myocardial infarction, etc. Orthotopic liver transplantation (OLT) is an effective treatment for that. Hepatocyte transplantation is an alternative to OLT that may help to overcome the shortage of donor organs. There have been reports of successful treatment of different kinds of metabolic liver disorders by hepatocyte transplantation. The major problem with hepatocyte transplantation is that the source of hepatocytes is very limited. Bone marrow stem cells are the potential source of hepatocytes. In the in-vitro culture system successful and efficient transdifferentiation of mesenchymal stem cells into hepatocytes has been documented. We have already shown that infusion of mesenchymal stem cells is safe and feasible in cirrhosis (Mohamadnejad M, et al. Arch Iran Med 2007; In Press). In this study, 2 patients with homozygous familial hypercholesterolemia will be included. The bone marrow of healthy volunteers with a normal lipid profile will be taken, then bone marrow mesenchymal stem cells (MSCs) will be cultured, and then MSCs will be trans-differentiate into hepatocytes, and the cells will be infused through the portal vein into the patients. The duration of follow up will be 6 months post-transplantation.

DETAILED DESCRIPTION:
Patients with homozygous familial hypercholesterolemia has very high serum cholesterol levels despite receiving lipid lowering drugs (e.g. statins, etc). Most of such patients die before the age of 20 due to myocardial infarction, etc. Orthotopic liver transplantation (OLT) is an effective treatment and can decrease their serum cholesterol to near normal levels (Bilheimer DW, N Engl J Med 1984; 311:1658-64). Shortage of donor organ is a major problem for OLT. Hepatocyte transplantation is an alternative to OLT that may help to overcome the shortage of donor organ. There have been reports of successful treatment of different kinds of metabolic liver disorders (such as Crigler Najjar Syndrome (Fox IJ, et al. N Engl J Med 1998;338:1422-6), Factor VII deficiency (Dhawan A et al. Transplantation 2004:78:1812-4), Glycogen storage disease type Ia (Muraca M, et al. Lancet 2002;359:317-8), etc) by hepatocyte transplantation. The major problem with hepatocyte transplantation is that the source of hepatocytes is very limited. Bone marrow stem cells are the potential source of hepatocytes. Although, in the in-vivo system there is a controversy that if stem cells transdifferentiate into hepatocytes or fusion of stem cells and hepatocytes occur, however, in the in-vitro culture system successful and efficient transdifferentiation of mesenchymal stem cells into hepatocytes has been documented (Lee KD, et al. Hepatology 2004;40:1275-1284; & Banas A, et al. Hepatology. 2007;46:219-28). We have already shown that infusion of mesenchymal stem cells is safe and feasible in cirrhosis (Mohamadnejad M, et al. Arch Iran Med 2007; In Press). In this study, 2 female patients with homozygous familial hypercholesterolemia will be included. The bone marrow of ABO compatible healthy male volunteers with a normal lipid profile will be taken, then bone marrow mesenchymal stem cells (MSCs) will be cultured, and then MSCs will be trans-differentiate into hepatocytes in the in-vitro culture system. Then the cells will be infused through the portal vein into the patients. The duration of follow up will be 6 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Severe hypercholesterolemia unresponsive to lipid lowering agents (e.g. statins)
* Presence of tendon xanthoma
* Documentation of homozygous familial hypercholesterolemia by appropriate genetic testing
* Female gender

Exclusion Criteria:

* Male gender

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Serum cholesterol and LDL levels | 6 Months

SECONDARY OUTCOMES:
Tracking the infused cells | Month 2 post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Digestive Disease Research Center, Medical Sciences/ Tehran University, Tehran, Iran; Hamid Goorabi, Phd, Study Chair — Royan Institute, Tehran, Iran; Mehdi Mohamadnejad, M.D., Principal Investigator — Digestive Disease Research Center, Medical Sciences/ Tehran University, Tehran, Iran; Hossein Baharvand, Phd, Principal Investigator — Department of Stem Cells, Royan Institute, Tehran, Iran
Locations (1):
- Digestive Disease Research Center, Shariati Hospital, North Kargar Ave., Tehran, Iran